CLINICAL TRIAL: NCT03041142
Title: Effects of an Interdisciplinary Intervention Program on Cardiovascular Risk Factors in Children With Overweight and Obesity
Brief Title: Program of Physical, Nutritional and Psychological Activities With Overweight Schoolchildren
Acronym: PANPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do vale do São Francisco (Other)
Responsible Party: Principal Investigator, THAYNA BEZERRA, Principal Investigator, Universidade Federal do vale do São Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 33
Record Dates: First submitted 2017-01-24; First posted 2017-02-02 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Cardiovascular Risk Factor
Keywords: Obesity; Cardiovascular risk factors; Interdisciplinary intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary Intervention (Experimental): Children 3 sessions/week 50-60 minutes of physical activity;
  1 session/week 60 minutes nutrition education week;
  1 session/week 120 minutes behaviour therapy.
  Mothers
  1 sessions/week 50-60 minutes of physical activity;
  1 session/week 60 minutes nutrition education week;
  1 session/week 120 minutes behaviour therapy.
  Interventions: Behavioral: Interdisciplinary intervention
- Routine (Active Comparator): Mothers and children followed their routine activities
  Interventions: Other: Routine

INTERVENTIONS:
Behavioral: Interdisciplinary intervention — Physical Activity, nutrition and Psychological
  Arms: Interdisciplinary Intervention
Other: Routine — The participants continued to maintain their routine
  Arms: Routine

SUMMARY:
Obesity has been considered as one of the primary factors for the development of pathologies and cardiovascular risk factors. In the child it has been mediator for the development of these comorbidities still in childhood, in the adolescence and more strongly in the adult age, at the time of most cardiovascular events with death records. Objective: To analyze the effects of an interdisciplinary intervention program on the cardiovascular risk factors of overweight and obese children. Methods: It was conducted a physical activity program, nutritional and psychological orientations, lasting ten weeks with overweighed children and their mothers. Thirty-three children with BMI considered overweight and obese participated in the study, they were divided into two groups, experimental (n=14) and control (n=19). Physical activities occurred 3 times a week with children and once a week with mothers. Nutritional and psychological counseling occurred once a week with both children and mothers. BMI, waist circumference, waist-height ratio, percentage of fat, cardiorespiratory fitness, systolic and diastolic blood pressure, lipid profile, glucose, left ventricular mass, daily energy intake and parental perception of children's weight were analyzed. For the statistical analysis it was first verified the normality of the data by the Shappiro Wilk test, with the variables that presented normality the possible differences were verified through the Anova test of mixed design with the post hoc of Bonferroni, for the normal variables, but that presented significant difference in the initial moment of the research, it was resorted to the Ancova, finally, for the non-normal variables the "U" tests of Mann Whitney and Wilcoxon.

DETAILED DESCRIPTION:
The intervention program was composed of physical activities, nutritional and psychological monitoring. The same lasted 10 weeks, where the meetings took place on Tuesdays and Thursdays with the children, in which they participated in 50 minutes of physical activity. On Saturdays, children were exposed to physical activity, guidance on healthy eating, and behavior change. On that day, mothers also participated in gym classes (duration of 50 minutes) and nutritional guidelines (duration of 50 minutes) and behavior change (duration of 120 minutes). It is noteworthy that the team was composed of ten psychology students and one teacher from the same area, three nutritionists, two teachers and five physical education students and four physicians.

Physical activities consisted of games and popular games lasting 50-60 minutes. Thus, in order to keep the children physically active as long as possible, timing was 2 minutes interval for water between each activity, resulting in a total time of 6 minutes rest throughout the class. Thus, there were 30 physical activity sessions with the children.

On Saturdays, mothers also participated in physical activities. Aerobic gymnastics and functional training were developed, lasting 50 minutes. During the classes, mothers were instructed to stay physically active during the week, performing, if possible, some physical activity at least five days a week.

On Saturdays, children were also submitted to guidelines on healthy eating, where they were encouraged to eat the right way, also learned about the importance of food, the group to which each food is a part, especially the foods they make Part of the context of the child, learned a variety of fruits and vegetables, learned how to prepare their own healthy snack and were motivated to take the acquired knowledge home, stimulating the whole family to adhere to healthier eating habits.

Nutrition counseling was also carried out with the mothers. At the meetings the nutritional needs for the age group of their children were exposed, the ideal foods to be consumed at each moment of the day, knowledge about the group to which each food belongs, adequate food According to the financial conditions, and a little book of recipes was created, where the food, fruits and typical dishes of the local region were emphasized, but in a healthier way.

Behavior change was stimulated by therapy with psychology trainees. The children were divided into 2 groups, to facilitate the process of psychological monitoring. The meetings were held once a week, on Saturdays, where activities and dynamics were developed with the aim of encouraging adherence to healthy habits, both food and physical activity. The therapies happened during 1 hour and they occurred in a playful way to involve all the universe of the child.

Mothers also had their moments of therapy, where they were motivated to be role models for their children, to stimulate this change in the children's lifestyle, they were also challenged to engage in some healthy activity during the week, at times alone, In others in the company of their children. Psychological encounters with mothers occurred on Saturdays, and they were divided into two groups to ensure greater control over the activities developed, as well as for them to feel more comfortable talking about themselves and their children. Parental relationships were extensively worked on in this practice. The meetings lasted two hours.

ELIGIBILITY:
Inclusion Criteria:

* Are regularly enrolled in municipal schools in the city of Petrolina-Pernambuco;
* They are classified as overweight or obese according to the criteria used by the researchers;
* Do not present restrictions to the practice of physical activities;
* Do not use medications that may interfere with your search results.

Exclusion Criteria:

* That they refuse to participate at some point in the data collection;
* That they have some restriction to the practices developed in the research, acquired during the course of the study;
* That they present a number greater than 50% of absences in the proposed activities;
* That parents or guardians miss four meetings or more.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-07-03 (Actual)

PRIMARY OUTCOMES:
Weight in kilograms | 5 minutes
  The weight was determined on Wiso® digital platform, model W801, with a precision of up to 100 g.
Height in meters | 5 minutes
  The stature was determined by means of a metal tape measure Sanny® attached to the wall, with precision of 0.1 cm.
Blood Pressure in millimeters of mercury | 20 minutes
  In order to measure blood pressure values among children, the Omron device (HEM 742) was used, consisting of an electronic and digital arm device, with inflation and automatic air deflation.
Lipid profile in milligrams per deciliter | 20 minutes
  For the dosages of the biochemical profile (triglycerides, total cholesterol, HDL-C and LDL-C) the blood was collected at the school itself by a nursing technique and the samples were taken to be analyzed in a specialized laboratory.
Left ventricular mass in grams | 30 minutes
  Transthoracic echocardiography was performed using the Vivid S6 echocardiogram model of the General Eletric® brand, year of manufacture 2011.

SECONDARY OUTCOMES:
Physical activity in minutes and bouts | 8 days.
  The level of physical activity was assessed using the Actigraph GT3X + accelerometer model (ActiGraph®, USA). The child wore the device at the waist for 8 days.
Sedentary behavior in minutes and bouts | 8 days
  The sedentary behavior was assessed using the Actigraph GT3X + accelerometer model (ActiGraph®, USA). The child wore the device at the waist for 8 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinando O Carvalho, Doctor, Study Director — Federal university of san francisco valley

IPD SHARING:
Plan to Share IPD: No